CLINICAL TRIAL: NCT05288569
Title: Immunological Biomarkers for Immune-related Adverse Events of Anti-PD-1/PD-L1 Immunotherapy in Lung Cancer: a Prediction Model
Brief Title: irAE Prediction of Anti-PD-1/L1 in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-2853
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Immune Checkpoint Inhibitors; Lung Cancer
Keywords: immunology; biomarkers; prediction; multidimensional
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and peripheral monocytes obtained from the peripheral blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the purpose of this study is to identify multi-dimensional immunological biomarkers including cytokines, autoantibodies, and immune cell subtypes of immune-related adverse events (primary) and prognosis(secondary) in the anti-PD-1/anti-PD-L1 immunotherapy for lung cancer

DETAILED DESCRIPTION:
After being informed of the study and potential risk, all patients giving written informed consent will undergo peripheral blood sample collection at baseline (before treatment ), 1month and 3month after treatment initiation, and when immune-related adverse events ever occur. The follow-up period will be 1 year for any occurrence of immune-related adverse events and 2 years follow-up for the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Stage I-IV Lung Cancer confirmed by histopathology or imaging techniques
* Receiving anti-PD-1/anti-PD-L1 immunotherapy (with indication and no contraindication)

Exclusion Criteria:

* Other cancer treatment
* Other malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at a national tertiary referral center for lung cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
occurrence of immune-related adverse event (irAE) | 12 months since immunotherapy initiation
  Any adverse events occured within 12 months since immunotherapy initiation will be independently evaluated by two clinicians to determine whether it is irAE and all the clinical characteristics of irAE will be documented

SECONDARY OUTCOMES:
Overall Survival | 24 months since immunotherapy initiation
  Patients will be followed up for 2 years to investigate Overall Survival
Progression Free Survival. | 24 months since immunotherapy initiation
  Patients will be followed up for 2 years to investigate Progression Free Survival.

CONTACTS AND LOCATIONS:
Overall Officials: Huaxia Yang, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Background] Yang H, Yao Z, Zhou X, Zhang W, Zhang X, Zhang F. Immune-related adverse events of checkpoint inhibitors: Insights into immunological dysregulation. Clin Immunol. 2020 Apr;213:108377. doi: 10.1016/j.clim.2020.108377. Epub 2020 Mar 2. PMID 32135278